CLINICAL TRIAL: NCT02140762
Title: A Phase 2b, Randomized, Controlled, Observer-Blind, Multi-Center Study Assessing the Effectiveness, Immunogenicity and Safety of Novartis Meningococcal ABCWY Vaccine Administered to Healthy Adolescents in the U.S.
Brief Title: Effectiveness, Immunogenicity and Safety of Meningococcal ABCWY Vaccine Administered to Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V102_16
Record Dates: First submitted 2014-05-06; First posted 2014-05-16 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Meningococcal Disease
Keywords: Meningitis ABCWY; Adolescents; Vaccination; Meningococcal disease
MeSH Terms: conditions — Meningococcal Infections | interventions — Saline Solution; MenACWY; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MenABCWY (Experimental): Subjects received one dose of MenABCWY vaccine at day 1 and a second dose after 2 months
  Interventions: Biological: MenABCWY
- Placebo/MenACWY (Active Comparator): Subjects received one dose of placebo at day 1 and one dose of MenACWY vaccine after 2 months
  Interventions: Other: Placebo; Biological: MenACWY

INTERVENTIONS:
Biological: MenABCWY — Subjects received one dose of 0.5 mL MenABCWY vaccine (intramuscular (IM) injection) at day 1 and a second dose after 2 months.
  Other Names: MenACWY conjugate combined with rMenB + OMV
  Arms: MenABCWY
Other: Placebo — 0.5 mL saline solution (IM)
  Other Names: saline solution
  Arms: Placebo/MenACWY
Biological: MenACWY — Subjects received one dose of 0.5 mL placebo (IM) at day 1 and one dose of 0.5 mL MenACWY vaccine (IM) after 2 months.
  Other Names: Menveo
  Arms: Placebo/MenACWY

SUMMARY:
Evaluate the effectiveness of 2 doses of MenABCWY vaccine in adolescents compared to a single dose of MenACWY vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents from 10-18 years of age, generally in good health, and available for all study visits, who/whose legally acceptable representative has given written informed consent at the time of enrollment.
* Female subjects of childbearing potential must have a negative urine pregnancy test.

Exclusion Criteria:

* Serious, acute, or chronic illnesses. Previous or suspected disease caused by N. meningitidis. Previous immunization with any meningococcal vaccine.
* Exposure to individuals with clinically proven meningococcal disease or clinical bacterial meningitis without further microbiologic characterization.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (8):
- United States (8):
  - Accelovance, Inc, Huntsville, Alabama
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Accelovance, Inc, Melbourne, Florida
  - Heartland Research Associates LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Meridian Clinical Research, Omaha, Nebraska
  - Senders Pediatrics, Cleveland, Ohio

REFERENCES:
- [Background] Adu-Bobie J, Capecchi B, Serruto D, Rappuoli R, Pizza M. Two years into reverse vaccinology. Vaccine. 2003 Jan 30;21(7-8):605-10. doi: 10.1016/s0264-410x(02)00566-2. PMID 12531326
- [Background] Bai X, Findlow J, Borrow R. Recombinant protein meningococcal serogroup B vaccine combined with outer membrane vesicles. Expert Opin Biol Ther. 2011 Jul;11(7):969-85. doi: 10.1517/14712598.2011.585965. Epub 2011 May 26. PMID 21615224
- [Derived] Viviani V, Biolchi A, Pizza M. Synergistic activity of antibodies in the multicomponent 4CMenB vaccine. Expert Rev Vaccines. 2022 May;21(5):645-658. doi: 10.1080/14760584.2022.2050697. Epub 2022 Mar 14. PMID 35257644
- [Derived] Welsch JA, Senders S, Essink B, Klein T, Smolenov I, Pedotti P, Barbi S, Verma B, Toneatto D. Breadth of coverage against a panel of 110 invasive disease isolates, immunogenicity and safety for 2 and 3 doses of an investigational MenABCWY vaccine in US adolescents - Results from a randomized, controlled, observer-blind phase II study. Vaccine. 2018 Aug 23;36(35):5309-5317. doi: 10.1016/j.vaccine.2018.07.016. Epub 2018 Jul 27. PMID 30061029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 8 study sites in USA.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenABCWY: Subjects received one dose of MenABCWY vaccine at visit day 1 and a second dose at visit month 2.
- Placebo/MenACWY: Subjects received one dose of placebo at visit day 1 and one dose of MenACWY vaccine at visit month 2.
Period: Overall Study
Arm/Group | MenABCWY | Placebo/MenACWY
Started | 154 | 151
Completed | 137 | 139
Not Completed | 17 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 9 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenABCWY | Placebo/MenACWY | Total
Number analyzed (Participants) | 154 | 151 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.9 (2.18) | 12.2 (2.42) | 12 (2.3)
Sex/Gender, Customized [Number; unit: participants]
  FEMALE | 67 | 61 | 128
  MALE | 87 | 90 | 177

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Without Bactericidal Activity at 1:4 Dilution Against Each US Neisseria Meningitidis (N. Meningitidis) Serogroup B Strain at One Month After the Second Vaccination.
Description: The combined percentage of subjects without bactericidal activity at 1:4 dilution using the endogenous complement human Serum Bactericidal Assay (enc-hSBA) across all strains in MenABCWY group and MenACWY group is reported at one month after the second injection. The percentage of subjects without bactericidal activity at 1:4 dilution was used to assess the effectiveness of two doses of MenABCWY vaccine when compared to one dose of Men ACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains.
  Least Square (LS)-mean computed from the generalized linear model.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on Full Analysis Set (FAS) effectiveness (month 3): all subjects in the All Enrolled Set who received a study vaccination and provided evaluable serum sample with enc-hSBA for at least one N. meningitidis serogroup B invasive disease strain at one month after the 2-dose series (Visit Month 3).
Measure: Mean (Standard Deviation); unit: Percentages of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 139 | 135
Percentages of subjects | 25.17 (30.77) | 76.19 (27.32)
Statistical Analysis 1: Comparison: MenABCWY vs Placebo/MenACWY; H0 (Null Hypothesis): Vaccine Effectiveness (VE) ≤10%. If the lower limit of the 95% CI for VE is > 10% the null hypothesis is to be rejected and effectiveness declared. The VE at 1 month after the 2nd injection for each strain is defined as [1-(% of subjects without bactericidal activity at 1:4 dilution in MenABCWY group / % of subjects without bactericidal activity at 1:4 dilution in MenACWY group)]x100. The combined VE across all strains will be computed by mean of a generalized linear model; Test type: Superiority or Other; p < 0.0001, Generalized Linear Model; Vaccine Effectiveness = 67, 95% CI 2-sided [65 to 69] — VE is based on the relative risk (RR). The Poisson Distribution and Log Link options were used in the generalized linear model to compute the log10 RR and the corresponding confidence interval. Fixed effects: treatment group, strain (and center)
Statistical Analysis 2: Comparison: MenABCWY vs Placebo/MenACWY; vaccine effectiveness<10% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity strains in ABCWY)/(% of not killed strains/without bactericidal activity strains in ACWY)*100]; Test type: Other — Vaccine effectiveness at one month after the second vaccination against each of the endemic US N.meningitidis serogroup B strains. Each individual strain data was analysed separately with treatment group as only independent variable in the model; Generalized Linear Model; Vaccine Effectiveness = 4.6
Statistical Analysis 3: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness <30% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity strains in ABCWY)/(% of not killed strains/without bactericidal activity strains in ACWY)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; generalized linear model; Vaccine Effectiveness = 12.7
Statistical Analysis 4: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<60% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity strains in ABCWY)/(% of not killed strains/without bactericidal activity strains in ACWY)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 18.2
Statistical Analysis 5: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness <100% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity strains in ABCWY)/(% of not killed strains/without bactericidal activity strains in ACWY)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 59.1

2. Secondary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:4 Dilution Against Each US N. Meningitidis Serogroup B Strain at 4 Months After the Second Vaccination.
Description: The combined percentage of subjects without bactericidal activity at 1:4 dilution using the endogenous complement human Serum Bactericidal Assay (enc-hSBA) across all strains in MenABCWY group and MenACWY group is reported at four months after the second injection. The percentage of subjects without bactericidal activity at 1:4 dilution was used to assess the effectiveness of two doses of MenABCWY vaccine when compared to one dose of Men ACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains.
  Least Square (LS)-mean computed from the generalized linear model.
Time Frame: Four months after the second vaccination (month 6)
Population: Analysis was done on FAS effectiveness (month 6): All subjects in the All Enrolled Set who received a study vaccination and provided evaluable serum sample with enc-hSBA for at least one N. meningitidis serogroup B invasive disease strain at four months after the 2-dose series (Visit Month 6).
Measure: Mean (Standard Deviation); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 136 | 135
Percentage of subjects | 42.91 (33.429) | 76.67 (27.706)
Statistical Analysis 1: Comparison: MenABCWY vs Placebo/MenACWY; H0 (Null Hypothesis): Vaccine Effectiveness (VE) ≤10%. If the LL of the 95% CI for VE is > 10% the null hypothesis is to be rejected and effectiveness declared. The VE at 4 months after the second injection for each strain is defined as [1 - (% of subjects without bactericidal activity at 1:4 dilution in MenABCWY group / % of subjects without bactericidal activity at 1:4 dilution in MenACWY group)] x 100.The combined VE across all strains will be computed by mean of a generalized linear model; Test type: Superiority or Other; p < 0.0001, General Linear Model (GLM); Vaccine effectiveness = 44, 95% CI 2-sided [41 to 47] — VE is based on the relative risk (RR). The POISSON DISTRIBUTION and LOG LINK options was used in the generalized linear model to compute the log10 RR and the corresponding confidence interval. Fixed effects: treatment group, strain (and center)
Statistical Analysis 2: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<10% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:4 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 9.1
Statistical Analysis 3: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<30% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:4 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 22.7
Statistical Analysis 4: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<60% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:4 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 19.1
Statistical Analysis 5: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<100% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:4 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 38.2

3. Secondary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:8 Dilution Against Each US N. Meningitidis Serogroup B Strain at One Month After the Second Vaccination
Description: The combined percentage of subjects without bactericidal activity at 1:8 dilution using the endogenous complement human Serum Bactericidal Assay (enc-hSBA) across all strains in MenABCWY group and MenACWY group is reported at one month after the second injection. The percentage of subjects without bactericidal activity at 1:8 dilution was used to assess the effectiveness of two doses of MenABCWY vaccine when compared to one dose of Men ACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains.
  Least Square (LS)-mean computed from the generalized linear model.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on FAS effectiveness ( month 3)
Measure: Mean (Standard Deviation); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 139 | 135
Percentage of subjects | 47.7 (37.04) | 88.28 (22.05)
Statistical Analysis 1: Comparison: MenABCWY vs Placebo/MenACWY; H0 (Null Hypothesis): Vaccine Effectiveness (VE) ≤ 10%. If the lower limit of the 95% CI for VE is >10% the null hypothesis is to be rejected and effectiveness declared. The VE at 1 month after the 2nd injection for each strain is defined as [1-(% of subjects without bactericidal activity at 1:8 dilution in MenABCWY group / % of subjects without bactericidal activity at 1:8 dilution in MenACWY group)]x100. The combined VE across all strains will be computed by mean of a generalized linear model; Test type: Superiority or Other; p < 0.0001, Generalized Linear Model; Vaccine Effectiveness = 46, 95% CI 2-sided [43 to 49] — VE is based on the relative risk (RR).The Poisson Distribution and Log Link options were used in the generalized linear model to compute the log10 RR and the corresponding confidence interval. Fixed effects:treatment group, strain (and center)
Statistical Analysis 2: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<10% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:8 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 25.5
Statistical Analysis 3: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<30%; Test type: Other — For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:8 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Vaccine Effectiveness = 19.1
Statistical Analysis 4: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<60% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:8 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 10.9
Statistical Analysis 5: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<100% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:8 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 40.9

4. Secondary Outcome: Percentages of Subjects Without Bactericidal Activity at 1:8 Dilution Against Each US N. Meningitidis Serogroup B Strain at Four Months After the Second Vaccination.
Description: The combined percentage of subjects without bactericidal activity at 1:8 dilution using the endogenous complement human Serum Bactericidal Assay (enc-hSBA) across all strains in MenABCWY group and MenACWY group is reported at four months after the second injection. The percentage of subjects without bactericidal activity at 1:8 dilution was used to assess the effectiveness of two doses of MenABCWY vaccine when compared to one dose of Men ACWY vaccine against a panel of US N. meningitidis serogroup B invasive disease strains.
  Least Square (LS)-mean computed from the generalized linear model.
Time Frame: Four months after the second vaccination (month 6)
Population: Analysis was done on FAS effectiveness (month 6).
Measure: Mean (Standard Deviation); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 136 | 135
Percentage of subjects | 70.89 (29.625) | 88.53 (21.442)
Statistical Analysis 1: Comparison: MenABCWY vs Placebo/MenACWY; H0 (Null Hypothesis): Vaccine Effectiveness (VE) ≤10%. If the lower limit of 95% CI for VE is > 10% the null hypothesis is to be rejected and effectiveness declared. The VE at 4 months after the 2nd injection for each strain is defined as [1 - (% of subjects without bactericidal activity at 1:8 dilution in MenABCWY group/% of subjects without bactericidal activity at 1:8 dilution in MenACWY group)] x 100. The combined VE across all strains was computed by mean of a generalized linear model; Test type: Superiority or Other; p < 0.0001, Generalized Linear Model — VE is based on the relative risk (RR). The POISSON DISTRIBUTION and LOG LINK options was used in the generalized linear model to compute the log10 RR and the corresponding confidence interval. Fixed effects: treatment group, strain (and center); Vaccine Effectiveness = 20, 95% CI 2-sided [16 to 23] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: MenABCWY vs Placebo/MenACWY; [analysis description as in outcome 3, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 36.4
Statistical Analysis 3: Comparison: MenABCWY vs Placebo/MenACWY; Vaccine effectiveness<30% For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated. For each strain, vaccine effectiveness (VE) of the MenABCWY compared to MenACWY was evaluated as VE= [1- (% not killed/without bactericidal activity at 1:8 dilution in MenABCWY group)/(% of not killed strains/without bactericidal activity in ACWY group)*100]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 15.5
Statistical Analysis 4: Comparison: MenABCWY vs Placebo/MenACWY; [analysis description as in outcome 3, analysis 4]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 20.9
Statistical Analysis 5: Comparison: MenABCWY vs Placebo/MenACWY; [analysis description as in outcome 3, analysis 5]; Test type: Other — [test comment as in outcome 1, analysis 2]; Vaccine Effectiveness = 11.8

5. Secondary Outcome: Percentages of N. Meningitidis Serogroup B Invasive Disease Strains Killed at 1:4 and 1:8 Dilutions, for Each Subject
Description: The mean percentage of N. meningitidis serogroup B invasive disease strains killed by each subject, at 1:4 and 1:8 dilutions at one month after the 2-dose vaccination series is reported.
Time Frame: Baseline, one month after second vaccination (month 3)
Population: Analysis was done on FAS effectiveness (month 3)
Measure: Mean (Standard Deviation); unit: Mean percentages of strains
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 139 | 135
Mean percentages of strains
  Baseline (1:4) (N=136, 132) | 20.08 (16.25) | 19.76 (15.48)
  1 month after 2nd vaccination (1:4) | 74.47 (14.55) | 22.93 (16.11)
  Baseline (1:8) (N=136, 132) | 9.25 (8.35) | 9.54 (9.49)
  1 month after 2nd vaccination (1:8) | 52.16 (17.11) | 11.39 (10.35)

6. Secondary Outcome: Percentages of N. Meningitidis Serogroup B Invasive Disease Strains Killed at 1:4 and 1:8 Dilutions, for Each Subject
Description: The mean percentage of N. meningitidis serogroup B invasive disease strains killed by each subject, at 1:4 and 1:8 dilutions at four months after the 2-dose vaccination series is reported.
Time Frame: Baseline, four months after second vaccination (month 6)
Population: Analysis was done on FAS effectiveness (month 6).
Measure: Mean (Standard Deviation); unit: Mean percentage of strains
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 136 | 135
Mean percentage of strains
  Baseline (1:4) (N=133, 132) | 19.82 (16.227) | 19.73 (15.079)
  4 months after 2nd vaccination (1:4) | 56.38 (18.703) | 22.66 (16.593)
  Baseline (1:8) (N=133, 132) | 9.19 (8.336) | 9.52 (9.346)
  4 months after 2nd vaccination (1:8) | 28.52 (18.484) | 11.19 (11.078)

7. Secondary Outcome: Percentages of Subjects With Enc-hSBA Titer >= 1:4 and Enc-hSBA Titer >= 1:8 at One Month After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY vaccine, in terms of percentages of subjects with enc-hSBA >= 1:4 and enc-hSBA titer >= 1:8 against four N. meningitidis serogroup B test strains at one month after the 2-dose vaccination series is reported.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on FAS Immunogenicity (Month 3): all subjects in the All Enrolled Set who received a study vaccination, provided evaluable serum samples respectively at 1 month post-second vaccination (Visit Month 3) whose immunogenicity assay result is available for at least one N. meningitidis serogroup B test strain or serogroups A, C, W or Y.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 134 | 130
Percentage of Subjects
  NZ98/254 (1:4, 1 month after 2nd vacc) (N=132,130) | 67 [57.9 to 74.6] | 1 [0.02 to 4.2]
  NZ98/254 (1:8, 1 month after 2nd vacc) (N=132,130) | 24 [17.2 to 32.5] | 0 [0 to 2.8]
  M14459 (1:4, 1 month after 2nd vacc) (N=134,129) | 96 [90.5 to 98.3] | 12 [7.3 to 19.4]
  M14459 (1:8, 1 month after 2nd vacc) (N=134,129) | 64 [55.4 to 72.3] | 3 [0.9 to 7.7]
  M07-0241084(1:4,1 month after 2nd vacc)(N=131,120) | 59 [49.8 to 67.3] | 20 [13.3 to 28.3]
  M07-0241084(1:8,1 month after 2nd vacc)(N=131,120) | 21 [14.7 to 29.4] | 7 [2.9 to 12.7]
  96217 (1:4, 1 month after 2nd vacc) (N=93,82) | 100 [96.1 to 100] | 49 [37.6 to 60.1]
  96217 (1:8, 1 month after 2nd vacc) (N=93,82) | 99 [94.2 to 99.97] | 15 [7.8 to 24.2]

8. Secondary Outcome: Percentages of Subjects With Enc-hSBA Titer ≥ 1:4 and Enc-hSBA Titer ≥ 1:8 at Four Months After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY vaccine, in terms of percentages of subjects with enc-hSBA ≥ 1:4 and enc-hSBA titer ≥ 1:8 against four N. meningitidis serogroup B test strains at four months after the 2-dose vaccination series is reported.
Time Frame: Four months after the second vaccination (month 6)
Population: Analysis was done on the FAS immunogenicity (month 6). The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 132 | 131
Percentage of subjects
  NZ98/254(1:4) (N=132,131) | 14 [8.9 to 21.6] | 5 [1.7 to 9.7]
  NZ98/254(1:8) (N=132,131) | 3 [0.8 to 7.6] | 2 [0.19 to 5.4]
  M14459 (1:4) (N=103,119) | 83 [73.8 to 89.3] | 20 [13.4 to 28.5]
  M14459(1:8) (N=103,119) | 26 [18 to 35.8] | 3 [0.5 to 7.2]
  M07-0241084 (1:4) (N=121,120) | 33 [24.8 to 42.2] | 19 [12.6 to 27.4]
  M07-0241084(1:8) (N=121,120) | 7 [3.5 to 13.7] | 7 [2.9 to 12.7]
  96217 (1:4) (N=87,76) | 100 [95.8 to 100] | 64 [52.7 to 75.1]
  96217 (1:8) (N=87,76) | 94 [87.1 to 98.1] | 14 [7.5 to 24.4]

9. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against the N. Meningitidis Serogroup B Test Strains
Description: The immunogenicity of two doses of MenABCWY compared to a single dose of MenACWY vaccine, in terms of hSBA GMTs against serogroup B test strains, at one month after the 2-dose vaccination series.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on FAS Immunogenicity (Month 3). The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 138 | 133
Titers
  NZ98/254 (1 month after 2nd vacc) | 6.03 [5.16 to 7.03] | 1.04 [0.89 to 1.22]
  M14459 (1 month after 2nd vacc) (N=138,132) | 13.4 [11 to 16] | 1.08 [0.92 to 1.28]
  M07-0241084 (1 month after 2nd vacc) (N=124,122) | 5.05 [4.08 to 6.26] | 1.65 [1.33 to 2.05]
  96217 (1 month after 2nd vacc) (N=124,118) | 169.22 [133 to 215] | 3.16 [2.48 to 4.04]

10. Secondary Outcome: HT-hSBA Geometric Mean Titers (GMTs) Against the N. Meningitidis Serogroup B Test Strains
Description: The immunogenicity of two doses of MenABCWY compared to a single dose of MenACWY vaccine, in terms of HT-hSBA GMTs against serogroup B test strains, at four months after the 2-dose vaccination series.
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 134
Titers
  NZ98/254 (N=133,134) | 1.75 [1.53 to 2] | 1.06 [0.93 to 1.21]
  M14459 (N=133,134) | 3.04 [2.6 to 3.56] | 1.12 [0.96 to 1.31]
  M07-0241084 (N=126,127) | 1.77 [1.47 to 2.12] | 1.56 [1.3 to 1.87]
  96217 (N=131,133) | 57.85 [45 to 74] | 3 [2.35 to 3.82]

11. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against the N. Meningitidis Serogroups A,C,W,Y
Description: The immunogenicity of two doses of MenABCWY compared to a single dose of MenACWY vaccine, in terms of hSBA GMTs to serogroups A, C, W, and Y, at one month after the 2-dose vaccination series.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on FAS Immunogenicity (Month 3)
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 137 | 125
Titers
  Men A (1 month after 2nd vacc) (N=137,115) | 77.02 [59 to 101] | 22.08 [17 to 30]
  Men C (1 month after 2nd vacc) (N=134,125) | 235.88 [171 to 325] | 38.61 [28 to 54]
  Men W (1 month after 2nd vacc) (N=119,115) | 157.72 [120 to 207] | 37.51 [28 to 49]
  Men Y (1 month after 2nd vacc) (N=107,94) | 155.43 [110 to 220] | 27.76 [19 to 40]

12. Secondary Outcome: HT-hSBA Geometric Mean Titers (GMTs) Against the N. Meningitidis Serogroups A, C, W, Y
Description: The immunogenicity of two doses of MenABCWY compared to a single dose of MenACWY vaccine, in terms of HT-hSBA GMTs to serogroups A, C, W, and Y, at four months after the 2-dose vaccination series.
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 133
Titers
  Men A (N=124,130) | 12.91 [9.19 to 18] | 5.56 [3.99 to 7.73]
  Men C (N=133,133) | 117.18 [84 to 163] | 25.64 [19 to 36]
  Men W (N=131,130) | 91.22 [70 to 119] | 42.97 [33 to 56]
  Men Y (N=132,132) | 59.51 [42 to 85] | 19.53 [14 to 28]

13. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against Serogroup B Test Strains ≥ Lower Limit of Quantitation (LLQ) at Baseline(Day 1) and One Month After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers against serogroup B test strains ≥ LLQ, at baseline(day 1) and one month after the 2-dose vaccination series, is reported. The LLQ cut off values for strains 96217, M07-0241084,M14459 and NZ98/254 were 8.6, 8.9, 8 and 8.2 respectively.
Time Frame: At baseline(day 1) and One month after the second vaccination (month 3)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 132 | 131
percentage of subjects
  96217 -Baseline (N=108,112) | 30 [21.2 to 39.2] | 32 [23.6 to 41.6]
  96217- Month 3 (N=119,114) | 99 [95.4 to 99.98] | 30 [21.6 to 39.1]
  M07-0241084-Baseline (N=123,128) | 3 [0.9 to 8.1] | 7 [3.3 to 12.9]
  M07-0241084-Month 3 (N=117,118) | 34 [25.7 to 43.5] | 10 [5.4 to 17.1]
  M14459-baseline(N=132,131) | 1 [0.02 to 4.2] | 1 [0.02 to 4.2]
  M14459-month 3 (N=131,128) | 73 [64.9 to 80.6] | 2 [0.49 to 6.7]
  NZ98/254-Baseline(N=131,131) | 1 [0.02 to 4.2] | 0 [0 to 2.8]
  NZ98/254-Month 3(N=131,129) | 44 [34.9 to 52.5] | 2 [0.19 to 5.5]

14. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroups A, C, W and Y ≥ LLQ at Baseline and One Month After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ against serogroups A, C, W, Y, at baseline(day 1) and one month after the 2-dose vaccination series.The LLQ cut off values for serogroups A,C,W and Y were 22.7,5.2,39.6 and 14.7 respectively.
Time Frame: At Baseline and One month after the second vaccination (month 3)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 130 | 131
percentage of subjects
  Men A -baseline(N=128,129) | 2 [0.19 to 5.5] | 1 [0.02 to 4.2]
  Men A- Month 3(N=130,112) | 93 [87.3 to 96.8] | 63 [52.9 to 71.5]
  Men C-baseline(N=130,131) | 32 [23.7 to 40.3] | 43 [34.2 to 51.7]
  Men C-Month 3(N=127,121) | 100 [97.1 to 100.0] | 82 [73.8 to 88.2]
  Men W-baseline(N=116,119) | 12 [6.8 to 19.4] | 16 [9.9 to 23.8]
  Men W-Month 3 (N=112,111) | 90 [83.1 to 95.0] | 52 [42.6 to 61.8]
  Men Y-baseline(N=122,123) | 10 [5.2 to 16.6] | 11 [5.8 to 17.4]
  Men Y-Month 3(N=102,91) | 96 [90.3 to 98.9] | 70 [59.8 to 79.5]

15. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against Serogroup B Test Strains ≥ Lower Limit of Quantitation (LLQ) at Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers against serogroup B test strains ≥ LLQ, at four months after the 2-dose vaccination series, is reported. The LLQ cut off values for strains 96217, M07-0241084,M14459 and NZ98/254 were 8.6, 8.9, 8 and 8.2 respectively
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 134
percentage of subjects
  96217 (N=131,133) | 95 [90.3 to 98.3] | 30 [22.4 to 38.6]
  M14459(N=133,134) | 26 [19.1 to 34.7] | 1 [0.18 to 5.3]
  M07-0231084 (N=126,127) | 10 [5.6 to 17.0] | 10 [5.6 to 16.9]
  NZ98/254(N=133,134) | 9 [4.8 to 15.2] | 1 [0.02 to 4.1]

16. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroups A, C, W and Y ≥ Lower Limit of Quantitation (LLQ) at Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ LLQ against serogroups A, C, W, Y at four months after the 2-dose vaccination series.The LLQ cut off values for serogroups A,C,W and Y were 22.7,5.2,39.6 and 14.7 respectively.
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 133
Percentages of subjects
  Men A (N=124, 130) | 48 [39.3 to 57.5] | 32 [24.4 to 41.1]
  Men C (N=133,133) | 98 [94.7 to 99.82] | 78 [70.2 to 84.9]
  Men W (N=131,130) | 77 [69.0 to 84.0] | 58 [48.7 to 66.3]
  Men Y (N=132,132) | 85 [77.6 to 90.5] | 63 [54.0 to 71.1]

17. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against Serogroup B Test Strains ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers against serogroup B test strains ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at four months after the 2-dose vaccination series, is reported.
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 134
Percentage of subjects
  NZ98/254 ≥ 5 (N=133,134) | 14 [8.8 to 21.4] | 2 [0.46 to 6.4]
  NZ98/254 ≥ 8 (N=133,134) | 9 [4.7 to 15.2] | 1 [0.18 to 5.3]
  NZ98/254 ≥ 16 (N=133,134) | 3 [0.8 to 7.5] | 0 [0 to 2.7]
  NZ98/254 ≥ 32 (N=133,134) | 2 [0.18 to 5.3] | 0 [0 to 2.7]
  NZ98/254 ≥ 64 (N=133,134) | 2 [0.18 to 5.3] | 0 [0 to 2.7]
  NZ98/254 ≥ 128 (N=133,134) | 1 [0.02 to 4.1] | 0 [0 to 2.7]
  M14459 ≥ 5 (N=133,134) | 39 [30.8 to 47.9] | 3 [0.8 to 7.5]
  M14459 ≥ 8 (N=133,134) | 26 [19.1 to 34.7] | 1 [0.18 to 5.3]
  M14459 ≥ 16 (N=133,134) | 9 [4.7 to 15.2] | 1 [0.02 to 4.1]
  M14459 ≥ 32 (N=133,134) | 2 [0.47 to 6.5] | 0 [0 to 2.7]
  M14459 ≥ 64 (N=133,134) | 1 [0.02 to 4.1] | 0 [0 to 2.7]
  M14459 ≥ 128 (N=133,134) | 0 [0 to 2.7] | 0 [0 to 2.7]
  M07-0241084 ≥ 5 (N=126,127) | 16 [10 to 23.4] | 13 [8 to 20.6]
  M07-0241084 ≥ 8 (N=126,127) | 11 [6.2 to 17.9] | 11 [6.2 to 17.8]
  M07-0241084 ≥ 16 (N=126,127) | 6 [2.3 to 11.1] | 8 [3.8 to 14]
  M07-0241084 ≥ 32 (N=126,127) | 2 [0.49 to 6.8] | 2 [0.19 to 5.6]
  M07-0241084 ≥ 64 (N=126,127) | 1 [0.02 to 4.3] | 0 [0 to 2.9]
  M07-0241084 ≥128 (N=126,127) | 0 [0 to 2.9] | 0 [0 to 2.9]
  96217 ≥ 5 (N=131,133) | 95 [90.3 to 98.3] | 35 [27.3 to 44.1]
  96217 ≥ 8 (N=131,133) | 95 [90.3 to 98.3] | 32 [23.8 to 40.2]
  96217 ≥ 16 (N=131,133) | 93 [87.4 to 96.8] | 22 [15.1 to 29.8]
  96217 ≥ 32 (N=131,133) | 77 [68.9 to 84] | 8 [3.7 to 13.4]
  96217 ≥ 64 (N=131,133) | 48 [39.3 to 57] | 5 [1.7 to 9.6]
  96217 ≥ 128 (N=131,133) | 19 [12.7 to 26.9] | 2 [0.18 to 5.3]

18. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroups A, C, W and Y ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at Four Months After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 against serogroups A, C, W, Y at four months after the 2-dose vaccination series.
Time Frame: Four months after the second vaccination (month 6)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- MenABCWY: Subjects received one dose of MenABCWY vaccine at visit day 1 and a second dose after visit month 2
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 133 | 133
Percentage of subjects
  Men A ≥ 8 (N=124,130) | 72 [63 to 79.5] | 43 [34.4 to 52]
  Men A ≥ 16 (N=124,130) | 65 [56.3 to 73.6] | 38 [29.3 to 46.6]
  Men A ≥ 32 (N=124,130) | 36 [27.8 to 45.4] | 29 [21.6 to 37.8]
  Men A ≥ 64 (N=124,130) | 16 [10.1 to 23.8] | 17 [10.9 to 24.5]
  Men A ≥ 128 (N=124,130) | 5 [1.8 to 10.2] | 8 [4.3 to 14.6]
  Men C ≥ 8 (N=133,133) | 97 [92.5 to 99.2] | 75 [67 to 82.3]
  Men C ≥ 16 (N=133,133) | 93 [87.5 to 96.9] | 55 [46 to 63.5]
  Men C ≥ 32 (N=133,133) | 82 [74.4 to 88.1] | 44 [35 to 52.5]
  Men C ≥ 64 (N=133,133) | 67 [58.2 to 74.8] | 32 [23.8 to 40.2]
  Men C ≥ 128 (N=133,133) | 47 [37.9 to 55.5] | 26 [18.4 to 33.8]
  Men W ≥ 8 (N=131,130) | 96 [91.3 to 98.7] | 87 [79.9 to 92.2]
  Men W ≥ 16 (N=131,130) | 95 [90.3 to 98.3] | 82 [74.6 to 88.4]
  Men W ≥ 32 (N=131,130) | 84 [76.5 to 89.8] | 66 [57.3 to 74.2]
  Men W ≥ 64 (N=131,130) | 61 [52.2 to 69.5] | 39 [30.8 to 48.2]
  Men W ≥ 128 (N=131,130) | 36 [27.7 to 44.7] | 24 [16.8 to 32.1]
  Men Y ≥ 8 (N=132,132) | 89 [82.8 to 94.1] | 67 [58.7 to 75.3]
  Men Y ≥ 16 (N=132,132) | 83 [75.9 to 89.3] | 61 [52.5 to 69.7]
  Men Y ≥ 32 (N=132,132) | 72 [63.5 to 79.4] | 48 [39.7 to 57.3]
  Men Y ≥ 64 (N=132,132) | 50 [41.2 to 58.8] | 37 [28.9 to 46]
  Men Y ≥ 128 (N=132,132) | 32 [24 to 40.5] | 19 [12.6 to 26.7]

19. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against Serogroup B Test Strains≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at One Month After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers against serogroup B test strains ≥ 5, ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at one month after the 2-dose vaccination series, is reported.
Time Frame: One month after the second vaccination (month 3)
Population: Analysis was done on the FAS immunogenicity (month 3). The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 138 | 133
Percentage of subjects
  NZ98/254 ≥ 5 (N=138,133) | 60 [51.5 to 68.4] | 2 [0.18 to 5.3]
  NZ98/254 ≥ 8 (N=138,133) | 45 [36.5 to 53.6] | 2 [0.18 to 5.3]
  NZ98/254 ≥ 16 (N=138,133) | 17 [11.5 to 24.8] | 0 [0 to 0.27]
  NZ98/254 ≥ 32 (N=138,133) | 5 [2.1 to 10.2] | 0 [0 to 2.7]
  NZ98/254 ≥ 64 (N=138,133) | 2 [0.45 to 6.2] | 0 [0 to 2.7]
  NZ98/254 ≥ 128 (N=138,133) | 1 [0.18 to 5.1] | 0 [0 to 2.7]
  M14459 ≥ 5 (N=138,132) | 83 [75.2 to 88.5] | 4 [1.2 to 8.6]
  M14459 ≥ 8 (N=138,132) | 73 [65 to 80.4] | 2 [0.47 to 6.5]
  M14459 ≥ 16 (N=138,132) | 56 [47.1 to 64.2] | 1 [0.02 to 4.1]
  M14459 ≥ 32 (N=138,132) | 22 [15.8 to 30.3] | 0 [0 to .28]
  M14459 ≥ 64 (N=138,132) | 7 [3.5 to 12.9] | 0 [0 to 2.8]
  M14459 ≥ 128 (N=138,132) | 0 [0 to 2.6] | 0 [0 to 2.8]
  M07-0241084 ≥ 5 (N=124,122) | 50 [40.9 to 59.1] | 16 [9.6 to 23.2]
  M07-0241084 ≥ 8 (N=124,122) | 40 [31.6 to 49.5] | 12 [7 to 19.5]
  M07-0241084 ≥ 16 (N=124,122) | 20 [13.5 to 28.3] | 7 [2.9 to 12.5]
  M07-0241084 ≥ 32 (N=124,122) | 5 [1.8 to 10.2] | 2 [0.5 to 7]
  M07-0241084 ≥ 64 (N=124,122) | 2 [0.5 to 6.9] | 1 [0.02 to 4.5]
  M07-0241084 ≥128 (N=124,122) | 2 [0.5 to 6.9] | 0 [0 to 3]
  96217 ≥ 5 (N=124,118) | 99 [95.6 to 99.98] | 34 [25.4 to 43.2]
  96217 ≥ 8 (N=124,118) | 99 [95.6 to 99.98] | 31 [23.1 to 40.5]
  96217 ≥ 16 (N=124,118) | 98 [94.3 to 99.8] | 21 [14.2 to 29.7]
  96217 ≥ 32 (N=124,118) | 96 [90.8 to 98.7] | 13 [7.3 to 20.1]
  96217 ≥ 64 (N=124,118) | 88 [80.8 to 93.1] | 4 [1.4 to 9.6]
  96217 ≥ 128 (N=124,118) | 66 [57.1 to 74.4] | 2 [0.21 to 6]

20. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers Against N. Meningitidis Serogroups A, C, W and Y ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128 at One Month After the 2-dose Vaccination Series
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with HT-hSBA titers ≥ 8, ≥ 16, ≥ 32, ≥ 64, ≥ 128, against serogroups A, C, W, Y, at one month after the 2-dose vaccination series.
Time Frame: One month after the second vaccination (month 3)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 137 | 125
Percentage of subjects
  Men A ≥ 8 (N=137,115) | 98 [93.7 to 99.55] | 72 [63 to 80.1]
  Men A ≥ 16 (N=137,115) | 96 [90.7 to 98.4] | 69 [59.4 to 77]
  Men A ≥ 32 (N=137,115) | 90 [83.4 to 94.3] | 57 [47.8 to 66.6]
  Men A ≥ 64 (N=137,115) | 66 [57.1 to 73.6] | 42 [32.6 to 51.3]
  Men A ≥ 128 (N=137,115) | 31 [23.7 to 39.9] | 19 [12.4 to 27.5]
  Men C ≥ 8 (N=134,125) | 99 [95.9 to 99.98] | 74 [65.8 to 81.8]
  Men C ≥ 16 (N=134,125) | 99 [95.9 to 99.98] | 64 [54.9 to 72.4]
  Men C ≥ 32 (N=134,125) | 98 [93.6 to 99.54] | 52 [42.9 to 61]
  Men C ≥ 64 (N=134,125) | 84 [77 to 90] | 39 [30.6 to 48.3]
  Men C ≥ 128 (N=134,125) | 68 [59.3 to 75.7] | 30 [22.5 to 39.3]
  Men W ≥ 8 (N=119,115) | 99 [95.4 to 99.98] | 86 [78.4 to 91.8]
  Men W ≥ 16 (N=119,115) | 98 [94.1 to 99.8] | 81 [72.5 to 87.6]
  Men W ≥ 32 (N=119,115) | 92 [85.1 to 95.9] | 61 [51.3 to 69.8]
  Men W ≥ 64 (N=119,115) | 79 [70.6 to 85.9] | 36 [26.9 to 45.1]
  Men W ≥ 128 (N=119,115) | 58 [48.6 to 67] | 23 [16.1 to 32.3]
  Men Y ≥ 8 (N=107,94) | 96 [90.7 to 99] | 71 [61 to 80.1]
  Men Y ≥ 16 (N=107,94) | 95 [89.4 to 98.5] | 69 [58.8 to 78.3]
  Men Y ≥ 32 (N=107,94) | 92 [84.6 to 96.1] | 63 [52.2 to 72.5]
  Men Y ≥ 64 (N=107,94) | 79 [70.5 to 86.6] | 48 [37.5 to 58.4]
  Men Y ≥ 128 (N=107,94) | 60 [49.9 to 69.2] | 30 [20.8 to 40.1]

21. Secondary Outcome: Percentage of Subjects With 2-fold Rise in hSBA Titer Against N.Meningitidis Serogroup B Strains at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a two-fold rise in HT-hSBA titers against the N.meningitidis serogroup B test strains, at 1 and 4 months after the 2-dose vaccination series.The 2-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥2 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 2 times of the prevaccination hSBA
Time Frame: At Month 3 and Month 6 ( one and four months after 2 doses of vaccination)
Population: Analysis was performed on FAS immunogenicity- month 3 and month 6. The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 137 | 131
Percentage of subjects
  96217-Month 3(N=101,99) | 92 [85.0 to 96.5] | 6 [2.3 to 12.7]
  M07-0241084-Month 3(N=115,119) | 13 [7.5 to 20.6] | 2 [0.20 to 5.9]
  M14459-Month 3(N=137,130) | 55 [46.8 to 64.0] | 0 [0 to 2.8]
  NZ98/254-Month 3(N=136,131) | 17 [11.0 to 24.3] | 0 [0 to 2.8]
  96217-Month 6(N=106,111) | 81 [72.4 to 88.1] | 5 [2.0 to 11.4]
  M07-0241084-Month 6(N=117,121) | 3 [0.5 to 7.3] | 1 [0.02 to 4.5]
  M14459-Month 6(N=132,131) | 9 [4.8 to 15.3] | 1 [0.02 to 4.2]
  NZ98/254-Month 6(N=131,131) | 2 [0.47 to 6.6] | 0 [0 to 2.8]

22. Secondary Outcome: Percentage of Subjects With 3-fold Rise in hSBA Titer Against N.Meningitidis Serogroup B Strains at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a 3-fold rise in HT-hSBA titers against the N.meningitidis serogroup B test strains, at 1 and 4 months after the 2-dose vaccination series.The 3-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥3 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 3 times of the prevaccination hSBA.
Time Frame: At Month 3 and Month 6 ( one and four months after 2 doses of vaccination)
Population: Analysis was performed on FAS immunogenicity-month 3 and month 6. The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 137 | 131
Percentage of subjects
  96217-month 3(N=101,99) | 91 [83.8 to 95.8] | 2 [0.25 to 7.1]
  M07-0231084-month 3(N=115,119) | 8 [3.6 to 14.3] | 0 [0 to 3]
  M14459-month 3(N=137,130) | 34 [26.4 to 42.9] | 0 [0 to 2.8]
  NZ98/254-month 3(N=136,131) | 10 [5.2 to 15.8] | 0 [0 to 2.8]
  96217-Month 6(N=106,111) | 70 [60.1 to 78.4] | 2 [0.22 to 6.4]
  M07-0241084-Month 6(N=117,121) | 2 [0.21 to 6.0] | 1 [0.02 to 4.5]
  M14459-Month 6(N=132,131) | 4 [1.2 to 8.6] | 0 [0 to 2.8]
  NZ98/254-Month 6(N=131,131) | 2 [0.47 to 6.6] | 0 [0 to 2.8]

23. Secondary Outcome: Percentage of Subjects With 4-fold Rise in hSBA Titer Against N.Meningitidis Serogroup B Strains at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a 4-fold rise in HT-hSBA titers against the N.meningitidis serogroup B test strains, at 1 and 4 months after the 2-dose vaccination series.
  The 4-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥4 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 4 times of the prevaccination hSBA.
Time Frame: At Month 3 and Month 6 ( one and four months after 2 doses of vaccination)
Population: Analaysis was performed on FAS immunogenicity-Month 3 and Month 6. The number of participants analyzed is the number of subjects assessed for this particular endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 137 | 131
Percentage of subjects
  96217-month 3(N=101,99) | 87 [79.0 to 93.0] | 1 [0.03 to 5.5]
  M07-0231084-month 3(N=115,119) | 2 [0.21 to 6.1] | 0 [0 to 3]
  M14459-month 3(N=137,130) | 22 [15.3 to 29.8] | 0 [0 to 2.8]
  NZ98/25-month 3(N=136,131) | 5 [2.1 to 10.3] | 0 [0 to 2.8]
  96217-Month 6(N=106,111) | 63 [53.3 to 72.4] | 1 [0.02 to 4.9]
  M07-0241084-Month 6(N=117,121) | 2 [0.21 to 6.0] | 0 [0 to 3]
  M14459-Month 6(N=132,131) | 2 [0.47 to 6.5] | 0 [0 to 2.8]
  NZ98/254-Month 6(N=131,131) | 2 [0.19 to 5.4] | 0 [0 to 2.8]

24. Secondary Outcome: Percentage of Subjects With 2-fold Rise in hSBA Titer Against N.Meningitidis Serogroups A,C,W and Y at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a two-fold rise in HT-hSBA titers against the N.meningitidis serogroups A,C,W and Y, at 1 and 4 months after the 2-dose vaccination series.
  The 2-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥2 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 2 times of the prevaccination hSBA.
Time Frame: At Month 3 and Month 6 ( one and four months after 2 doses of vaccination)
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 132 | 130
Percentage of subjects
  Men A-month 3(N=132,110) | 81 [73.3 to 87.4] | 48 [38.6 to 57.9]
  Men C-month 3(N=131,123) | 98 [94.6 to 99.81] | 66 [56.8 to 74.2]
  Men W-month 3(N=107,103) | 74 [64.5 to 81.9] | 25 [17.2 to 34.8]
  Men Y-Month 3(N=99,86) | 92 [84.7 to 96.5] | 59 [48.2 to 69.8]
  Men A-Month 6(N=119,126) | 23 [15.5 to 31.3] | 21 [13.9 to 28.8]
  Men C-Month 6(N=130,130) | 94 [88.2 to 97.3] | 55 [45.7 to 63.4]
  Men W-Month 6(N=114,116) | 54 [43.9 to 62.9] | 30 [22.0 to 39.4]
  Men Y-Month 6(N=122,121) | 72 [63.3 to 79.9] | 47 [38.0 to 56.4]

25. Secondary Outcome: Percentage of Subjects With 3-fold Rise in hSBA Titer Against N.Meningitidis Serogroups A, C, W and Y at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a three-fold rise in HT-hSBA titers against the N.meningitidis serogroups A,C,W and Y at 1 and 4 months after the 2-dose vaccination series.
  The 3-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥3 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 3 times of the prevaccination hSBA.
Time Frame: At Month 3 and Month 6 (one and four months after 2 doses of vaccination)
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 132 | 130
Percentage of subjects
  Men A-Month 6(N=119,126) | 13 [7.9 to 20.9] | 14 [8.7 to 21.6]
  Men C-Month 6(N=130,130) | 88 [81.7 to 93.4] | 48 [38.9 to 56.6]
  Men W-Month 6(N=114,116) | 32 [24.0 to 41.9] | 22 [14.5 to 30.2]
  Men Y-Month 6(N=122,121) | 61 [51.4 to 69.4] | 40 [31.7 to 49.8]
  Men A-Month 3(N=132,110) | 61 [51.7 to 69.0] | 36 [27.4 to 46.1]
  Men C-Month 3(N=131,123) | 98 [94.6 to 99.81] | 58 [48.5 to 66.6]
  Men W-Month 3(N=107,103) | 56 [46.2 to 65.7] | 19 [12.3 to 28.4]
  Men Y-Month 3(N=99,86) | 85 [76.2 to 91.3] | 50 [39.0 to 61.0]

26. Secondary Outcome: Percentage of Subjects With 4-fold Rise in hSBA Titer Against N.Meningitidis Serogroups A,C,W and Y at One and Four Months After the 2-dose Vaccination Series.
Description: The immunogenicity of two doses of MenABCWY vaccine compared to a single dose of MenACWY, in terms of the percentages of subjects with a 4-fold rise in HT-hSBA titers against the N.meningitidis serogroups A,C,W and Y, at 1 and 4 months after the 2-dose vaccination series.
  The 4-fold rise in titer is defined as follows:
  a)for subjects with prevaccination hSBA titers <LLQ, a postvaccination hSBA ≥4 LLQ; b) for subjects with a prevaccination hSBA titers ≥LLQ, an increase of at least 4 times of the prevaccination hSBA.
Time Frame: At Month 3 and Month 6 ( one and four months after 2 doses of vaccination)
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 132 | 130
Percentage of subjects
  Men A-Month 3(N=132,110) | 45 [36.0 to 53.6] | 26 [18.4 to 35.6]
  Men C-month 3(N=131,123) | 95 [89.3 to 97.8] | 54 [44.4 to 62.7]
  Men W-Month 3(N=107,103) | 50 [39.7 to 59.4] | 15 [8.4 to 22.9]
  Men Y-month 3(N=99,86) | 81 [71.7 to 88.0] | 47 [35.7 to 57.6]
  Men A-Month 6(N=119,126) | 8 [3.5 to 13.9] | 11 [6.2 to 17.9]
  Men C-Month 6(N=130,130) | 86 [79.0 to 91.6] | 43 [34.4 to 52.1]
  Men W-Month 6(N=114,116) | 27 [19.3 to 36.3] | 17 [10.9 to 25.4]
  Men Y-Month 6(N=122,121) | 49 [40.0 to 58.4] | 35 [26.3 to 43.9]

27. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Reactogenicity was presented in terms of number of subjects reporting solicited local and systemic AEs and other indicators.
Time Frame: From day 1 (6 hours) until day 7 after any vaccination
Population: Analysis was done on Solicited Safety Set: all subjects in the All Exposed Set who have provided any solicited adverse event data and/or other indicators or reactogenicity
Measure: Number; unit: subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 149 | 146
subjects
  Any | 129 | 92
  Any Local Reactions | 128 | 65
  Any Systemic Reactions | 70 | 66
  Induration (mm) (N=149,145) | 21 | 8
  Erythema (mm) (N=149,145) | 23 | 5
  Pain (N=149,145) | 127 | 63
  Nausea | 9 | 19
  Fatigue | 40 | 35
  Myalgia | 20 | 14
  Arthralgia | 18 | 5
  Headache | 40 | 42
  Fever (N=148,146) | 9 | 0
  Chills | 15 | 8
  Loss of appetite | 23 | 12
  Prevention of pain/fever (N=149,144) | 4 | 2
  Treatment of pain/fever (N=149,144) | 60 | 9

28. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs.
Description: Percentages of subjects reporting unsolicited AEs including serious adverse events (SAEs).
Time Frame: From day 1 to day 30 after any vaccination for any unsolicited AE. From day 1 to study termination (day 181) for all other categories.
Population: Analysis was done on the unsolicited safety set, ie, all subjects in the exposed set with any unsolicited adverse event data and/or indicators of unsolicited adverse events. Analysis for AEs leading to withdrawal was done on All Enrolled Set population.
Measure: Number; unit: Subjects
Arm/Group | MenABCWY | Placebo/MenACWY
Number analyzed (Participants) | 150 | 146
Subjects
  Any unsolicited AEs | 28 | 28
  Possibly or probably related AEs | 7 | 3
  Medically-attended AEs | 37 | 44
  AEs leading to withdrawal | 1 | 1
  Any SAEs | 0 | 1
  SAE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs): from Day 1 to Day 7 of each study vaccination. Unsolicited AEs from Day 1 to Day 30 after each vaccination. Serious AEs, medically attended AEs, AEs leading to withdrawal were collected for the whole duration of the study.
Description: Data are presented in terms of number of subjects reporting AEs and in terms of number of subjects reporting AEs with a frequency >5% in at least one group. For serious AEs, analysis was done on Unsolicited Safety set. For solicited/unsolicited AEs with a frequency >5%, analysis was done on Overall Safety Set.
Arm/Group | MenABCWY | Placebo/MenACWY
All-Cause Mortality (participants affected / at risk) | 0/150 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/150 | 1/146
Other Adverse Events (participants affected / at risk) | 132/151 | 100/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenABCWY (N=150) | Placebo/MenACWY (N=146)
PHARYNGITIS (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenABCWY (N=151) | Placebo/MenACWY (N=147)
NAUSEA (Gastrointestinal disorders) | 10 | 20
CHILLS (General disorders) | 15 | 9
FATIGUE (General disorders) | 42 | 40
INJECTION SITE ERYTHEMA (General disorders) | 60 | 24
INJECTION SITE INDURATION (General disorders) | 51 | 16
INJECTION SITE PAIN (General disorders) | 130 | 71
PYREXIA (General disorders) | 11 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 19 | 7
MYALGIA (Musculoskeletal and connective tissue disorders) | 23 | 15
HEADACHE (Nervous system disorders) | 42 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No